CLINICAL TRIAL: NCT05997589
Title: Money Matters 101: A Pilot Community-Based Financial Health Educational Program
Brief Title: Financial Health Educational Program for Increasing Financial Literacy Among Underserved Communities in Western New York
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I 3445122; NCI-2023-02314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 3445122 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Behavior Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (educational program) (Experimental): Participants attend financial health educational program over 60 minutes. Patients also receive educational materials on study.
  Interventions: Behavioral: Behavioral Intervention; Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive educational materials
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Educational Intervention — Attend financial health educational program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a financial health educational program to educate and increase knowledge for financial health and well-being, and to ensure access to financial knowledge and resources among underserved community members in Western New York. Financial well-being consists of a person's ability to meet financial obligations, feelings of financial security, ability to make choices related to financial matters. Information gathered from this study may help researchers learn how a financial health educational program may increase financial literacy for financial health and well-being among underserved community members in Western New York.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collaborate with community organizations and leaders to leverage community-based assets to disseminate education about financial literacy.

II. Reach medically underserved, high risk community members. III. Enhance financial literacy knowledge among medically underserved, high risk community members.

OUTLINE:

Participants attend financial health educational program over 60 minutes. Patients also receive educational materials on study.

After completion of study intervention, patients are followed up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old

Exclusion Criteria:

* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Success of program dissemination (Feasibility) | Up to 1 year
  Will be measured by number and demographics of attendees at each programs offered organizations to deliver financial health literacy education. Descriptive statistics will be used to summarize demographic and baseline characteristics.
Satisfaction of financial health educational program (Acceptability) | Up to 1 year
  Descriptive statistics will be used to summarize demographic and baseline characteristics.
Effectiveness of community based education | Up to 1 year
  Demographics of attendees at each program will determine the effectiveness of this community-based educational strategy to reach diverse, high-risk, and medically underserved community members.

SECONDARY OUTCOMES:
Changes in financial literacy knowledge | Baseline to 1 year
  Will use surveys to collect questionnaire data before and after education sessions. Scores from the pre- and post-knowledge tests will be computed as the average percent correct of the responses to each question and then will be compared across all participants. Comparisons of pre-post test scores will be made using paired-samples t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States